CLINICAL TRIAL: NCT03727698
Title: Prospective Evaluation of Radiotherapy Using Magnetic Resonance Image Guided Treatment
Acronym: PERMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4841
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: To assess delivery of radiotherapy on the MR Linac for multiple tumour sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy delivered on the MR Linac (Experimental): MR Guided radiotherapy treatment
  Interventions: Device: MR Linac

INTERVENTIONS:
Device: MR Linac — MR guided radiotherapy treatment

SUMMARY:
The purpose of PERMIT is to collect information on the treatment of radiotherapy patients using a new radiotherapy machine that includes magnetic Resonance (MR) imaging (MR linac) to guide treatment. The aim is to use this information to support the introduction of MR Linac into clinical practice.

PERMIT will collect details on patients treated on the MR linac plus details on their side effects and other outcomes. This information plus technical and imaging information will be combined with information from other centres using this machine. By doing so this will help us learn how best to use the MR Linac in the future and design new radiotherapy protocols

ELIGIBILITY:
Inclusion Criteria:

1. Radiotherapy treatment suitable to be delivered on the MR Linac.
2. Patient provides written, informed consent and/or authorization.
3. Patients between the ages of 5 and under 16 years old may enter protocol with parental/guardian consent.

Exclusion Criteria:

1. Contra-indications to MR imaging.
2. Radiotherapy not suitable for delivery on the MR Linac e.g. those with extended field lengths (exceeding 20 cm).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Technical feasibility of undertaking MRL based radiotherapy at multiple clinical sites: The percentage of treatment fractions delivered successfully on the MR linac | 2 years
  The percentage of treatment fractions delivered successfully on the MR linac, if more than 20 % of patients (depending on treatment site) need to be treated on alternative machine or treatment protocol changed will lead to the MRL protocol at that site to be judged not feasible.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHSFT, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared within the academic and industrial partners. All data sharing would be dependant on appropriate data sharing agreements.
Supporting Information: Study Protocol, SAP, CSR